CLINICAL TRIAL: NCT04195321
Title: Norepinephrine Versus Phenylephrine Infusion for Prophylaxis Against Spinal Induced Hypotension in Elderly Undergoing Hip Arthroplasty Under Spinal Anesthesia: A Randomized Comparative Trial
Brief Title: Norepinephrine Versus Phenylephrine for Preventing Spinal Anesthesia Induced Hypotension in Elderly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Maha Mostafa Ahmad, MD, Principal Investigator, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D-7-2019
Record Dates: First submitted 2019-12-06; First posted 2019-12-11 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Spinal Induced Hypotension; Elderly
MeSH Terms: interventions — Norepinephrine; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- norepinephrine group (Active Comparator): patients will receive NE infusion at a starting of rate of 1 ml/min of 8 mcg/ml solution (prepared by diluting 4 mg NE in 500 ml normal)
  Interventions: Drug: Norepinephrine
- phenylephrine (Active Comparator): patients will receive PE infusion at a starting rate of 1 ml/min of 100 mcg/ml solution (prepared by diluting 10 mg of PE in 100 ml normal saline)
  Interventions: Drug: phenylephrine

INTERVENTIONS:
Drug: Norepinephrine — infusion will be started after induction of spinal anesthesia
  Arms: norepinephrine group
Drug: phenylephrine — infusion will be started after induction of spinal anesthesia
  Arms: phenylephrine

SUMMARY:
Various regimens were used for prevention of hypotension; most of these regimens included the use of vasopressors. Ephedrine is commonly used vasopressor for management and prophylaxis of hypotension; however, ephedrine is usually associated with tachycardia which increases oxygen consumption; thus, it might be potentially harmful in this special group of patients. Phenylephrine (PE) is another vasopressor which is characterized by α agonistic activity. PE had been the preferred vasopressor for prophylaxis against post-spinal hypotension especially in obstetric population.

it was reported that PE improved the intraoperative hemodynamic profile in elderly patients undergoing lower extremities orthopedic surgery under spinal anesthesia. PE (a pure α agonist) was reported to decrease cardiac output which limit its use in patients with compromised cardiac contractility; this fact makes the use of PE in elderly patients questionable. Norepinephrine (NE) is characterized by α agonistic and weak β agonistic activity; thus, NE is characterized by less cardiac depression compared to PE. NE was recently introduced for prophylaxis against post-spinal hypotension in obstetric anesthesia. In non-obstetric population, although, NE infusion effectively maintained patients hemodynamics during general anesthesia, its use during spinal anesthesia was not adequately evaluated in elderly population

DETAILED DESCRIPTION:
Preoperative fasting instructions are 6 hours for solid food, and clear fluid will be allowed up to 2 hours preoperative. Upon arrival to the operating room, routine monitors (ECG, pulse oximetry, and non-invasive blood pressure monitor) will be applied; intravenous line will be secured, and routine pre-medications (ranitidine 50 mg and midazolam 0.02 mg/kg slow IV) will be administrated. Baseline preoperative blood pressure will be recorded in the supine position as average of 3 reading with difference less than 5 mmHg.

Fluid management:

Before initiation of spinal anesthesia for all study patients, Electrical cardiometry device (ICON; Cardiotonic, Osypka; Berlin, Germany) will be applied to the patient through 4 electrodes at the following sites: Below the left ear, Above the midpoint of the left clavicle, Left mid-axillary line at level of the xiphoid process and 5 cm inferior to the third electrode. Stroke volume variability (SVV) will be measured while patient maintaining standard calm breathing at a rate of 6-8 breath/minute before the intrathecal injection. The patient with SVV more than 13% with be considered fluid responder 16 and will receive fluid bolus of 5 ml/kg ringer acetate over 10 minutes. The fluid bolus will be repeated till SVV less than 13%, then spinal anesthesia will be performed. After induction of spinal anesthesia maintenance fluid as 2ml/kg/hour of ringer acetate will be commenced.

Anesthetic management:

Spinal anesthesia will be performed in the sitting position at level of second and third or third and forth lumber interspaces with a 25-gauge spinal needle. After confirming cerebrospinal fluid flow, 10 mg of 0.5% hyperbaric bupivacaine plus 25 mcg fentanyl will be injected. The degree of sensory block (cold test by alcohol gauze) will be assessed in the study with a goal of T6-8 dermatomal level block. If spinal anesthesia failed, the patient will be excluded from the study and will be managed according to the attending anesthetist discretion, local expertise and clinical practice.

Vasopressor management:

Vasopressor infusion will be started after obtaining CSF through the same line with IV fluids aided by a three-way stop-cock after induction of spinal anesthesia, patients will receive the vasopressor infusion according to the previous randomization Any episode of spinal induced hypotension (defined as mean arterial pressure < 80% of the baseline reading 30 minutes after spinal block) will be managed by 5 mcg norepinephrine and the infusion rate will be increased by 20%. If the hypotensive episode persisted for 2 minutes, another bolus of norepinephrine will be administered.

If bradycardia (defined as heart rate less than 50 bpm) with hypotension occurred, it will be manged with 0.5 mg of atropine IV. If bradycardia occurred with hypertension (MAP increase 25% over the baseline), the vasopressor infusion will be stopped.

If hypertension occurred (defined as increased mean arterial pressure by > 25% of the baseline reading), vasopressor infusion will be decreased by 50%. If hypertension persisted 2 minutes after reduction of the infusion, the vasopressor infusion will be stopped. The vasopressor will be returned to 50% of the starting dose if there was further decline in blood pressure.

The infusion will continue for 45 minutes after spinal anesthesia. If the patient developed hypotension after stoppage of the infusion, management will depend on the fluid status of the patient. If the cause of hypotension was blood loss, replacement will be done (3:1 of ringer acetate till transfusion threshold met then packed RBC is given with target haemoglobin ≥9gm/dl). If the hypotension was not related to blood loss, vasopressor will be re-initiated at the last dose before stoppage

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients (>65), ASA I-II-III, scheduled for hip joint surgery under spinal anesthesia

Exclusion Criteria:

* Contraindication of spinal anesthesia (patient's refusal, infection at injection site, allergy, increased intracranial tension, coagulopathy, tight valvular lesion),
* history of allergy to any of the study's drugs,
* Patients with cardiac morbidities (impaired contractility with ejection fraction < 50%, heart block, arrhythmias),
* hypertensive patients,
* patients on beta blockers,
* patient with hyperthyroidism
* patients on monoamine oxidase inhibitors (MAOI) will be excluded from the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
mean heart rate | for 45 minutes starting 2 minutes after induction of spinal anesthesia
  beat per minute

SECONDARY OUTCOMES:
incidence of bradycardia | for 45 minutes starting 2 minutes after induction of spinal anesthesia
  heart rate less than 60 beat per minute
incidence of reactive hypertension | for 45 minutes starting 2 minutes after induction of spinal anesthesia
  increased mean arterial pressure by > 25% of the baseline reading
Incidence of spinal induced hypotension | for 45 minutes starting 2 minutes after induction of spinal anesthesia
  mean arterial pressure < 80% of the baseline reading 45 minutes after induction of spinal anesthesia and not related to blood loss

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alaini Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided